CLINICAL TRIAL: NCT04427254
Title: Study of the Sars-Cov2 Neuroinvasiveness - COVID19
Acronym: CORONEVRAXE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment number not reached
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBN_2020_16
Record Dates: First submitted 2020-05-26; First posted 2020-06-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: COVID19
Keywords: Sars-Cov2 neuroinvasiveness; COVID-19 RT-PCR test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurological biological samples (Experimental)
  Interventions: Drug: Cerebrospinal fluid sampling, meningeal and brain parenchyma biopsies

INTERVENTIONS:
Drug: Cerebrospinal fluid sampling, meningeal and brain parenchyma biopsies — Cerebrospinal fluid sampling, meningeal and brain parenchyma biopsies

SUMMARY:
Sars-Cov2 (COVID-19) may invade the CNS inducing neurological diseases such as anosmia, ageusia, encephalitis, ischemic or hemorrhagic stroke. Management of severe neurological complications in COVID-19 patients may require ventricular cerebrospinal fluid drainage and cranial decompression. During surgery, cerebrospinal fluid, meninges and brain parenchyma can be safely removed from the patient. In this study, COVID-19 patients will be evaluated first, for the presence of Sars-Cov2 in the cerebrospinal fluid and/or biopsies and second, for the consequences of Sars-Cov2 neuroinfection in terms of inflammatory and immune responses.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients requiring an external ventricular drain, a decompressive craniectomy or an intracranial hematoma surgery

Exclusion Criteria:

* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with COVID-19 positive samples/biopsies | At the time of the inclusion
  COVID-19 RT-PCR test

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOURDILLON, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A de Rothschild, Paris, France